CLINICAL TRIAL: NCT06630247
Title: A Dose-escalation, Dose-finding, and Expansion Study of XL495 as a Single Agent and in Combination Therapy in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Dose-escalation, Dose-finding, and Expansion Study of XL495 in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XL495-101
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Solid Cancers; Solid Tumor Cancer; Solid Tumor Malignancy; Urothelial Cancer (Urinary Bladder, Ureters, or Renal Pelvis Cancer); Metastatic Solid Tumor; Locally Advanced Solid Tumor; Urothelial Cancer of Renal Pelvis
Keywords: solid tumor; renal tumor; metastatic solid tumor; urothelial carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Renal Cell; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: This study is divided into three stages:
  The first stage is the dose escalation stage that evaluates how much of XL495 alone patients can safely tolerate.
  The second is the dose finding stage that evaluates how much of XL495 to give patients in combination with other anti-cancer medications.
  The third stage is the expansion stage that evaluates how XL495 performs in patients in combination with other anti-cancer medications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation XL495 (Experimental): Group(s) of participants with advanced metastatic tumors who will receive increasing doses of XL495.
  Interventions: Drug: XL495
- Dose Finding XL495 + ADC cytotoxic agents (Experimental): Group(s) of participants with advanced metastatic tumors who will receive XL495 and Antibody drug conjugate (ADC) cytotoxic agents together at increasing doses.
  Interventions: Drug: XL495; Drug: ADC cytotoxic agents
- Expansion XL495 + ADC cytotoxic agents (Experimental): Group(s) of participants with urothelial cancer who will receive XL495 and ADC cytotoxic agents at the recommended dosage(s) of expansion (RDE [s]) determined during the dose-escalation and dose-finding stages.
  Interventions: Drug: XL495; Drug: ADC cytotoxic agents

INTERVENTIONS:
Drug: XL495 — oral doses of XL495
Drug: ADC cytotoxic agents — intravenous infusion of anti-cancer combination agent
  Arms: Dose Finding XL495 + ADC cytotoxic agents; Expansion XL495 + ADC cytotoxic agents

SUMMARY:
The goal of this study is to obtain safety, tolerability, PK, and preliminary clinical antitumor activity for XL495 as a single agent and in combination with select cytotoxic agents in participants with locally advanced or metastatic tumors for whom life-prolonging therapies do not exist or available therapies are intolerable/no longer effective.

ELIGIBILITY:
Inclusion Criteria

* For All Participants

  * Have received at least one standard therapy unless it does not exist, or available therapies are intolerable or no longer effective.
  * For participants, who qualify for approved molecularly selected therapies such as RAS inhibitors, they must have progressed on, relapsed from, been intolerant to, ineligible, or refused those therapies.
* Expansion Stage

  * Diagnosis of metastatic advanced UC (primary tumor: renal pelvis, ureter, urinary bladder, or urethra).
  * At least one measurable lesion as defined by RECIST, version 1.1.
  * Participants must be eligible for sacituzumab govitecan treatment as their next line of therapy.
* At least one but no more than 3 prior lines of therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (0-2 for monotherapy; 0-1 for combo)

Exclusion Criteria

* Prior anticancer treatment, including:

  * Radiation therapy within 2 weeks before first dose of study treatment.
* Known brain metastases or cranial epidural disease
* Current or recent severe illness
* Known history or positive test for human immunodeficiency virus (HIV) unless meets specific criteria.
* Active infection with hepatitis B virus or hepatitis C virus.
* Malabsorption syndrome.
* History of solid organ, autologous or allogenic stem cell transplant.
* Diagnosis of another cancer within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with standard therapy.
* Active autoimmune disease with skin involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Dose-escalation and Dose-finding Stages: Number of Participants with Treatment-Emergent Adverse Events | Up to 18 months
Dose-escalation and Dose-finding Stages: Number of Participants with Dose-limiting Toxicities | Up to 18 months
Expansion Stage: Number of Participants with Treatment-Emergent Adverse Events | Up to 19 months
Expansion Stage: Objective Response Rate (ORR) As Assessed by Investigator Per RECIST 1.1 | Until disease progression or death, up to approximately 19 months
  ORR is defined as the percentage of participants with the best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), as assessed by the Investigator per RECIST 1.1.

SECONDARY OUTCOMES:
Dose-escalation and Dose-finding Stages: Concentration of XL495 in Plasma | Pre-dose and multiple post-dose time points, up to 18 months
Dose-escalation and Dose-finding Stages: Pharmacokinetic (PK) Parameter Area Under the Plasma Concentration Time Curve (AUC) of XL495 | Pre-dose and multiple post-dose time points, up to 18 months
Dose-escalation and Dose-finding Stages: PK Parameter Maximum Plasma Concentration of XL495 (Cmax) | Pre-dose and multiple post-dose time points, up to 18 months
Dose-escalation and Dose-finding Stages: PK Parameter Time to Cmax of XL495 (Tmax) | Pre-dose and multiple post-dose time points, up to 18 months
Dose-escalation and Dose-finding Stages: PK Parameter Apparent Clearance with Oral Administration of XL495 (CL/F) | Pre-dose and multiple post-dose time points, up to 18 months
Dose-escalation and Dose-finding Stages: PK Parameter Apparent Terminal Elimination Half-life of XL495 (t1/2) | Pre-dose and multiple post-dose time points, up to 18 months
Expansion Stage: Duration of Response (DOR) As Assessed by Investigator per RECIST 1.1 | Until disease progression or death, up to approximately 19 months.
  DOR is defined as the time from the first documented objective response (CR or PR) until the earlier of radiographic progressive disease (PD) as assessed by the investigator per RECIST 1.1 or censoring due to lack of these events or start of non-protocol anti-cancer therapy.
Expansion Stage: Progression-free Survival (PFS), as Assessed by Investigator per RECIST 1.1 | Until disease progression or death, up to approximately 19 months.
  PFS is defined as the time from start of study treatment to the earlier of either radiographic PD per RECIST 1.1 or death from any cause.
Expansion Stage: Concentration of XL495 in Plasma | Pre-dose and multiple post-dose time points, up to 18 months
Expansion Stage: Pharmacokinetic (PK) Parameter Area Under the Plasma Concentration Time Curve (AUC) of XL495 | Pre-dose and multiple post-dose time points, up to 18 months
Expansion Stage: PK Parameter Maximum Plasma Concentration of XL495 (Cmax) | Pre-dose and multiple post-dose time points, up to 18 months
Expansion Stage: PK Parameter Time to Cmax of XL495 (Tmax) | Pre-dose and multiple post-dose time points, up to 18 months
Expansion Stage: PK Parameter Apparent Clearance with Oral Administration of XL495 (CL/F) | Pre-dose and multiple post-dose time points, up to 18 months
Expansion Stage: PK Parameter Apparent Terminal Elimination Half-life of XL495 (t1/2) | Pre-dose and multiple post-dose time points, up to 18 months

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Exelixis Clinical Site #4, Denver, Colorado
  - Exelixis Clinical Site #9, New Haven, Connecticut
  - Exelixis Clinical Site #8, Washington D.C., District of Columbia
  - Exelixis Clinical Site #10, Jefferson, Louisiana
  - Exelixis Clinical Site #7, New York, New York
  - Exelixis Clinical SIte #2, Huntersville, North Carolina
  - Exelixis Clinical Site #3, Nashville, Tennessee
  - Exelixis Clinical Site #5, Nashville, Tennessee
  - Exelixis Clinical Site #1, Austin, Texas
  - Exelixis Clinical Site #6, Houston, Texas